CLINICAL TRIAL: NCT01279213
Title: Augmentation of Clozapine With Paliperidone in the Treatment of Resistant Schizophrenia Randomized Controlled Study
Brief Title: Clozapine/Paliperidone Versus Clozapine/Placebo in Resistant Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: DANIEL SERRANI, faculty of psychology UNR
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 109
Record Dates: First submitted 2011-01-11; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-07

CONDITIONS: Schizophrenia; Schizophrenic Disorders; Psychotic Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paliperidone clozapine BPRS (Active Comparator): patients assigned to clozapine plus paliperidone controls at 6 and 12 weeks
  Interventions: Drug: paliperidone clozapine
- clozapine plus placebo BPRS (Placebo Comparator): patients assigned to placebo plus clozapine should show less improvement
  Interventions: Drug: paliperidone clozapine

INTERVENTIONS:
Drug: paliperidone clozapine — dose 3 to 12 mg paliperidone ER daily during 12 weeks

SUMMARY:
augmentation of clozapine with paliperidone in the treatment of resistant schizophrenia has not been tested until now in randomized controlled trials. This combination is supposed to have therapeutic efficacy in the treatment of resistant schizophrenia.

DETAILED DESCRIPTION:
This is a 12 weeks, blind study (the patient, investigator, and sponsor do not know the study drug and dosage being taken by the patient) of the safety and tolerability of flexible-dose (3 to 12mg per day), extended-release (ER) paliperidone in combination with clozapine with a diagnosis of schizophrenia. Patients who have completed study or who discontinued from that study because of lack of efficacy but completed a minimum of 21 days of the study may enter this study. This study consists of a 21-day screening and washout phase (to discontinue and "wash out" any medication not allowed in the study), and a double blind treatment phase of 12 weeks, during which all patients will take oral paliperidone ER every day and clozapine versus clozapine alone, and a post-treatment phase consisting of a follow-up visit completed 1 week after a patient has received the final dose of paliperidone ER. The study, including the screening and posttreatment phase, will last approximately 30 weeks. Screening and washout may be conducted while a patient is an outpatient. Safety will be assessed by laboratory measurements (chemistry, liver function tests, hematology, hormone, lipid assessments, prolactin [blinded], urinalysis, and urine drug screens; body weight, height, and waist circumference measurements; ECGs and the ESRS (extrapyramidal syndrome rating scale). These instruments will be used to assess extrapyramidal symptoms (EPS) and dyskinesias. Adverse events will be monitored including psychiatric adverse events of interest (worsening of psychosis, hyperprolactinemia, weight gain) that may be associated with paliperidone ER in this population. The primary aim of this study is to evaluate the long-term (12 weeks) safety and tolerability of clozapine/paliperidone ER in resistant schizophrenia. As exploratory secondary aims, the study will assess the effect of clozapine/paliperidone ER on the long-term symptoms of schizophrenia as measured by the changes in the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scores, the global improvement in severity of illness as measured by the Clinical Global Impression(CGI) scale. Patients begin the study at 6.0 mg/day of oral paliperidone ER. If a higher dosage is needed, the dosage will be increased (in increments of 3 mg/day not more frequently than once every 5 days) to 12 mg/day. If the 6.0 mg/day dosage is not well tolerated, the dosage may be decreased (not more frequently than once every 5 days) to 3.0 mg/day. Patients will be dosed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

resistant schizophrenia failure in therapeutic response to three previous antipsychotic drugs -

Exclusion Criteria:

age upper 50 other psychiatric diagnosis head trauma neurological diseases -

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
bprs | 12 weeks
  improvement in scores total BPRS

SECONDARY OUTCOMES:
cgs | 12 weeks
  improvement in CGS

CONTACTS AND LOCATIONS:
Overall Officials: daniel j serrani azcurra, MD, Principal Investigator — faculty of psychology
Locations (1):
- Faculty of Psychology, Rosario, Santa Fe Province, Argentina

REFERENCES:
- [Background] Mortimer AM, Singh P, Shepherd CJ, Puthiryackal J. Clozapine for treatment-resistant schizophrenia: National Institute of Clinical Excellence (NICE) guidance in the real world. Clin Schizophr Relat Psychoses. 2010 Apr;4(1):49-55. PMID 20643629